CLINICAL TRIAL: NCT06914310
Title: Memantine as an Additive Therapy in Patients With Traumatic Brain Injury
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Noha Mansour, Associate professor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-88
Record Dates: First submitted 2025-03-27; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Mild Traumatic Brain Injury; Moderate Traumatic Brain Injury (TBI)
Keywords: Traumatic Brain Injury (TBI); Memantine; S100β
MeSH Terms: conditions — Brain Concussion; Brain Injuries, Traumatic | interventions — Memantine; Mannitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Memantine group (Active Comparator): Mild to moderate TBI patients will receive memantine. It will be given either orally or through a nasogastric tube for 7 days, starting on the first day of admission to the hospital and then continued for 3 weeks. The memantine dose in the first 7 days is 30 mg twice daily, while during the remaining 3 weeks the dose is 10 mg twice daily
  Interventions: Drug: Memantine
- Control group (Other): Mild to moderate TBI patients will be managed by mannitol or hypertonic saline to reduce brain swelling and analgesic for headache such as; acetaminophen.
  Interventions: Drug: Mannitol

INTERVENTIONS:
Drug: Memantine — Memantine will be given either orally or through a nasogastric tube for 7 days, starting on the first day of admission to the hospital and then continued for 3 weeks. The memantine dose in the first 7 days is 30 mg twice daily, while during the remaining 3 weeks the dose is 10 mg twice daily
  Arms: Memantine group
Drug: Mannitol — Mild to moderate TBI patients will receive mannitol in case of brain edema to reduce brain swelling and analgesic for headache such as; acetaminophen.
  Arms: Control group

SUMMARY:
Memantine has shown promise in mitigating secondary brain injury in previous studies. One study demonstrated that early memantine administration in moderate TBI patients resulted in lower serum neuron-specific enolase levels and improved Glasgow Coma Scale scores. However, other trials investigating memantine's impact on long-term cognitive function in TBI patients have yielded mixed results. There is a need for well-controlled studies to determine the efficacy of memantine in improving neurological and cognitive outcomes in patients with TBI.

DETAILED DESCRIPTION:
The current study aims to evaluate the cognitive function, neuroprotective effect, and S-100β serum level effect of Memantine in patients with mild to moderate traumatic brain injury (TBI) patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 18 and 70 years of age
2. Patients mild (GCS 13-15) to moderate (GCS 9-12) TBI were assessed for the study eligibility.

Exclusion Criteria:

1. Comorbid illnesses, such as diabetes mellitus, ischemic heart disease, acute myocardial infarction within the past 48 hours.
2. Acute or chronic renal insufficiency.
3. Hepatic diseases.
4. Autoimmune diseases.
5. Malignancies.
6. Pregnancy.
7. Patients unable to tolerate enteral feeding.
8. More than 24 hours (h) since traumatic injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-25 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
The difference between the 2 groups regarding mean Montreal Cognitive Assessment (MOCA) scores at the end of treatment | 30 days
  Score rage: 0 - 30. Normal cognition: 26 - 30, mild cognitive impairment: 18 - 25, moderate cognitive impairment: 10 - 17 and severe cognitive impairment: less than 10.

SECONDARY OUTCOMES:
The differences between study groups in Glasgow Coma Scale (GCS) score. | 3 days
  The differences between study groups in GCS scores over 3 days. The score ranges from 3 (Minimum score = deep coma or death) to 15 (Maximum score = fully awake and oriented). Traumatic brain injury (TBI) is graded as mild, moderate, or severe on the basis of the level of consciousness or Glasgow coma scale (GCS) score after resuscitation. Mild TBI score ranges from 13 to 15, moderate TBI ranges from 9 to 13; while severe TBI ranges from 3 to 8.
The difference between the two study groups in mean serum level of S100 calcium-binding protein B (S100B) | 3 days
  The difference between the two study groups in mean serum level of S100 calcium-binding protein B (S100B) .

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No